CLINICAL TRIAL: NCT03445897
Title: Miltefosine Combined With Intralesional Pentamidine for Leishmania Braziliensis Cutaneous Leishmaniasis in Bolivia
Brief Title: Miltefosine Plus IL Pentamidine for Bolivian CL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jonathan Berman (Other)
Responsible Party: Sponsor-Investigator, Jonathan Berman, President, AB Foundation
Organization: AB Foundation (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABF MP
Record Dates: First submitted 2018-02-21; First posted 2018-02-26 (Actual); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Leishmaniasis, Cutaneous
MeSH Terms: conditions — Leishmaniasis, Cutaneous | interventions — miltefosine

STUDY DESIGN:
Intervention Model Description: Bolivian cutaneous leishmaniasis due to Leishmania braziliensis was treated with the combination of miltefosine (150 mg/day for 28 days) plus intralesional pentamidine (120 ug/mm2 lesion area on days 1, 3, and 5).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): miltefosine (150 mg/day for 28 days) plus intralesional pentamidine (120 ug/mm2 lesion area on days 1, 3, and 5).
  Interventions: Drug: miltefosine plus intralesional pentamidine

INTERVENTIONS:
Drug: miltefosine plus intralesional pentamidine — miltefosine (150 mg/day for 28 days) plus intralesional pentamidine (120 ug/mm2 lesion area on days 1, 3, and 5).

SUMMARY:
Bolivian cutaneous leishmaniasis due to Leishmania braziliensis was treated with the combination of miltefosine (150 mg/day for 28 days) plus intralesional pentamidine (120 ug/mm2 lesion area on days 1, 3, and 5).

DETAILED DESCRIPTION:
Bolivian cutaneous leishmaniasis due to Leishmania braziliensis was treated with the combination of miltefosine (150 mg/day for 28 days) plus intralesional pentamidine (120 ug/mm2 lesion area on days 1, 3, and 5). Efficacy and tolerance parameters were assessed. Efficacy was assessed at 1, 3, and 6 months post therapy. Tolerance was assessed on each day therapy was administered.

ELIGIBILITY:
Inclusion Criteria:

* one ulcerative lesion ≤ 900 mm2 in total area,
* ≥ 12 years,
* parasitologically diagnosed by visualization of amastigotes or culture of promastigotes from lesion material,
* no antileishmanial therapy in the last 3 months,
* no mucosal lesions,
* no history of significant concomitant diseases including immunosuppression.

Exclusion Criteria:

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-01-31 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-02-21 (Actual)

PRIMARY OUTCOMES:
Lesion size | 6 months post therapy
  area of lesion

SECONDARY OUTCOMES:
adverse effects at site | days 1, 3, 5 of therapy
  pain, erythema, edema
systemic adverse effects | days 1 to 28 of therapy
  gastrointestinal side effects

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2015-10-05): https://cdn.clinicaltrials.gov/large-docs/97/NCT03445897/Prot_000.pdf